CLINICAL TRIAL: NCT02715752
Title: A Retrospective Chart Review Study of Gene-Eden-VIR/Novirin
Status: Completed | Type: Observational
Sponsor: The Center for the Biology of Chronic Disease (Other)
Responsible Party: Sponsor
Other Study IDs: 022015
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Herpes Simplex Infections; Human Papillomavirus; Epstein-Barr Virus Infections; Varicella-zoster Virus Infection; Cytomegalovirus Infections
MeSH Terms: conditions — Herpes Simplex; Epstein-Barr Virus Infections; Varicella Zoster Virus Infection; Cytomegalovirus Infections | interventions — Gene-Eden-VIR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Herpes Simplex Virus Infection: Gene-Eden-VIR/Novirin, oral, 1-4 capsules per day, 12 months
  Interventions: Dietary Supplement: Gene-Eden-VIR/Novirin
- Human Papillomavirus Infection: Gene-Eden-VIR/Novirin, oral, 1-4 capsules per day, 12 months
  Interventions: Dietary Supplement: Gene-Eden-VIR/Novirin
- Epstein-Barr Virus Infection: Gene-Eden-VIR/Novirin, oral, 1-4 capsules per day, 12 months
  Interventions: Dietary Supplement: Gene-Eden-VIR/Novirin
- Cytomegalovirus Infection: Gene-Eden-VIR/Novirin, oral, 1-4 capsules per day, 12 months
  Interventions: Dietary Supplement: Gene-Eden-VIR/Novirin
- Varicella Zoster Virus Infection: Gene-Eden-VIR/Novirin, oral, 1-4 capsules per day, 12 months
  Interventions: Dietary Supplement: Gene-Eden-VIR/Novirin

INTERVENTIONS:
Dietary Supplement: Gene-Eden-VIR/Novirin

SUMMARY:
This study measured the changes in health-related complaints by analyzing charts of individuals, who are infected with a latent virus, who have used Gene-Eden-VIR/Novirin.

DETAILED DESCRIPTION:
The medical community calls the movement from severe to mild disease and from mild to normal health, 'relieving symptoms', and the interventions that cause such movement, drugs, medications, or therapies. The alternative community calls the movement from normal health to superior health, 'boosting health' (or boosting the immune system, or improving your sex drive, or boosting any another well functioning physiological system), and the interventions that cause such movement, natural remedies, dietary supplements, complementary treatments, etc. In general, these interventions aim to achieve superior performance of a normal human body. Of course, boosting the body's normal performance improves many of its capabilities, such as higher resistance to diseases, faster recovery from fatigue, better mental concentration, etc. Each movement presents different objectives. Relieving symptoms represents the ability of an intervention to reduce the frequency, duration, and severity of a disease. In contrast, boosting health represents the ability of an intervention to increase the frequency, duration, and quality of a person's health. In the current study, the investigators would like to measure the changes in health-related complaints by analyzing charts of individuals, who are infected with latent virus, and who have used Gene-Eden-VIR/Novirin.

ELIGIBILITY:
Inclusion Criteria:

* Latent viral infection with either HSV, HPV, VZV, EBV, or CMV
* Taking Gene-Eden-VIR/Novirin

Exclusion Criteria:

* Use of other antiviral treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women ages greater than 18 years old
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
frequency of symptoms | one year
duration of symptoms | one year

SECONDARY OUTCOMES:
time to first recurrence | one year

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for the Biology of Chronic Disease, Valley Cottage, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Polansky H, Itzkovitz E, Javaherian A. Clinical study of Gene-Eden-VIR/Novirin in genital herpes: suppressive treatment safely decreases the duration of outbreaks in both severe and mild cases. Clin Transl Med. 2016 Dec;5(1):40. doi: 10.1186/s40169-016-0121-6. Epub 2016 Oct 20. PMID 27766602